CLINICAL TRIAL: NCT07183891
Title: Head-to-Head Evaluation of ChatGPT 4o, GPT-5, and DeepSeek for Structured Extraction, Toric IOL Recommendation, and Refractive Prediction
Brief Title: Performance of Large Language Models for Structured Recognition and Refractive Prediction
Status: Recruiting | Type: Observational
Sponsor: Jin Yang (Other)
Responsible Party: Sponsor-Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Other Study IDs: Totic-2025-001
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cataract
Keywords: cataract; toric IOL; astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We conducted a single-center, retrospective observational study to evaluate large language models (ChatGPT 4o, GPT-5, DeepSeek) for automated interpretation of de-identified IOLMaster 700 reports provided as raster images. Models produced structured biometric extraction, toric IOL recommendation, and refractive predictions (sphere, cylinder, axis). Primary outcomes included parameter-level agreement and refractive error metrics; secondary outcomes included decision-support performance for toric IOL selection and agreement on ordered T-codes. No clinical intervention was performed.

DETAILED DESCRIPTION:
This study compares three large language models accessed in their native configurations, without fine-tuning or external tools. For each examination, the original IOLMaster 700 report image was supplied without manual annotation or pre-processing. A standardized instruction required: (i) structured extraction of AL, ACD, LT, WTW, K1/K2 and axes, ΔK, TK1/TK2 and axes, and ΔTK; (ii) binary toric candidacy and T-code according to institutional ALCON mapping; and (iii) refractive recommendations (sphere, cylinder, implantation axis). Each model generated three independent outputs per case. De-identification and IRB oversight (waiver of consent) were implemented according to institutional policy. The unit of enrollment is participants (n=54), with outcomes analyzed per eye (162 eyes) and per model generation where applicable.

ELIGIBILITY:
Inclusion Criteria:

-postoperative corrected distance visual acuity (CDVA) of 0.10 logMAR or better -an absolute IOL rotational stability of less than 10∘ at the 1-month follow-up examination

Exclusion Criteria:

* incomplete biometric data on the examination report;
* a history of previous ocular surgery or ocular trauma
* the occurrence of intraoperative complications, such as an anterior capsular tear or posterior capsular rupture
* the development of significant postoperative complications, including but not limited to severe intraocular infection or inadequate pupillary dilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cataract patients who had undergone phacoemulsification and implantation of an AcrySof IQ Toric monofocal intraocular lens
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Refractive prediction error for sphere | At index examination
  Mean absolute error (MAE, diopters) of model-predicted sphere versus clinical reference
Cohen's kappa with 95% CIs between model | At index examination (single time point)
  Cohen's kappa with 95% CIs between model outputs and clinician-validated reference for per-parameter

SECONDARY OUTCOMES:
Cylinder prediction error | At index examination
  Mean absolute error (MAE, diopters) of model-predicted Cylinder
Axis prediction error | At index examination
  Mean absolute error (MAE, diopters) of model-predicted Axis

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No